CLINICAL TRIAL: NCT03188055
Title: Best Case/Worst Case Trauma Study: A Communication Tool to Assist Severely Injured Older Adults
Brief Title: A Communication Tool to Assist Severely Injured Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Oregon Health and Science University (Other); University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2016-1588; R21AG055876-01 (NIH)
Record Dates: First submitted 2017-06-12; First posted 2017-06-15 (Actual); Results first posted 2020-12-28 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2020-12

CONDITIONS: Communication
Keywords: patient decision making; surgical decision making; shared decision making; decision support techniques
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best Case/Worst Case communication tool (Experimental): The patient's enrolled surgeon will have completed training on the Best Case/Worst Case communication tool and will be encouraged to use it with the patient.
  Interventions: Other: Best Case/Worst Case communication tool
- Usual Care (No Intervention): Usual care typically includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention.Usual care also consists of daily updates with patient and family, describing each new problem as it arises and what will be done to treat it, regardless of how this fits into the patient's overall prognosis or health trajectory.

INTERVENTIONS:
Other: Best Case/Worst Case communication tool — The communication tool promotes dialogue and patient deliberation, and supports shared decision making in the context of life-limiting illness. Building on a conceptual model of shared decision-making proposed and the practice of scenario planning our intervention is designed to lead to a discussion of patient preferences and consideration of outcomes.
  The surgeon verbally describes the "best case," "worst case," and "most likely" outcomes for each treatment option-incorporating rich narrative from clinical experience and translation of probabilistic information-while drawing a diagram of those options. The surgeon also writes details about each option on the diagram. The narrative and graphic help family and patients formulate and express preferences.
  Arms: Best Case/Worst Case communication tool

SUMMARY:
The purpose of this study is to test the effect of the "Best Case/Worse Case" (BC/WC) communication tool on the quality of communication with older patients admitted to two trauma units. The intervention was developed and tested with acute care surgical patients at the University of Wisconsin (UW) and we are now testing whether the intervention will work in a different setting. We will test the intervention with severely injured older adults at Oregon Health Sciences University (OHSU) and Parkland Memorial Hospital (PMH) at the University of Texas Southwestern (UTS). In the first year, UTS/PMH and OHSU will recruit and enroll 50 patients in the control arm (total, for both sites) and train trauma surgeons to use the best case/worst case tool. In the second year, UTS/PMH and OHSU will recruit and enroll 50 patients in the intervention arm (total, for both sites). UW will compare survey-reported and chart-derived measures before and after clinicians learn to use the best case/worst case tool.

DETAILED DESCRIPTION:
The purpose of this study is to test the effect of the "best case/worse case" communication tool on the quality of communication with older patients admitted to two trauma units and to collect feedback on the tool to help adapt it to the trauma setting. The intervention was developed and tested with acute care surgical patients at the University of Wisconsin (UW) and the present study seeks to test whether the intervention will work in a different setting.

To adapt the tool to trauma settings, we will conduct focus groups at UW Health Oregon Health Sciences University (OHSU) and Parkland Memorial Hospital (PMH) at the University of Texas-Southwestern (UT-S). Because trauma care is delivered by a multidisciplinary team, we will include attending trauma surgeons, surgical residents, ICU nurses, nurse practitioners, consulting physicians (e.g. orthopedic surgeons) and others on the trauma care team. Up to 60 trauma car providers will participate in focus groups across the three sites. We will test the intervention with severely injured older adults at OHSU and UT-S/PMH. In the first year, UT-S/PMH and OHSU will recruit and enroll 50 patients total in the control arm and train trauma surgeons to use the best case/worst case tool. In the second year, UT-S/PMH and OHSU will recruit and enroll 50 patients total in the intervention arm.

UT-S/PMH and OHSU research team members will survey family members of trauma patients to compare the quality of communication for severely injured geriatric trauma patients cared for by trauma teams. When possible, UT-S/PMH and OHSU will survey patients on their quality of life. UT-S/PMH and OHSU will survey the patient's primary nurse on the quality of communication patients and will survey patient's families about their thoughts on the quality of communication as well. UT-S/PMH and OHSU will survey trauma unit staff before and after clinicians learn to use the best case/worst case tool, to assess whether the communication intervention improves feelings of moral distress. UT-S/PMH and OHSU will use chart review to collect downstream clinical outcomes including intensity of treatment and receipt of palliative care. UT-S/PMH and OHSU will archive de-identified graphic aids used by trauma surgeons with intervention patients to explore how the intervention was enacted.

ELIGIBILITY:
Patients

Inclusion Criteria:

* Traumatically injured patients 50 and older admitted to the ICU

Exclusion Criteria:

* Surgeons will have an opportunity to exclude a patient or family who, in the physician's judgment, would not be an appropriate participant
* Patients with a Physician Orders for Life-Sustaining Medical Treatment (POLST) or Medical Orders for Life-Sustaining Medical Treatment (MOLST) form on file in their medical record that specifies that the patient or their decision maker wishes them to receive no intervention
* Patients with an isolated head injury as defined by a Head Abbreviated Injury Scale (AIS) score of 2 or less and an External AIS score of 1 or 0 and a Glasgow Coma Scale (GCS) score of 15. This serves to exclude the mildly traumatically brain injured patients with minimal external injuries who require ICU-level monitoring for a short period of time only

Family Members

Inclusion Criteria:

* N/A

Exclusion Criteria:

* We will exclude patients whose family members do not speak English
* Under the age of 18
* Lack decision making capacity (DMC)
* Have a severe hearing or vision impairment.

Surgeons

Inclusion Criteria:

-N/A

Exclusion Criteria:

* Care providers who do not directly provide primary trauma care in the ICU
* Residents who have not had at least 5 years of postgraduate training
* Trauma consultants including for example, neurosurgeons, orthopedic surgeons, and otolaryngologists

Nurses

Inclusion Criteria:

* The nurse responsible for care of the enrolled patient at 3 days post-admission will be invited to complete a Quality of Communication (QOC) survey assessment

Exclusion Criteria:

* N/A

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Schwarze, MD, MPP, FACS, Principal Investigator — University of Wisconsin, Madison; Karen Brasel, MD, MPH, Principal Investigator — Oregon Health and Science University; Thomas Shoultz, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (2):
- United States (2):
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas Southwestern, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zimmermann CJ, Zelenski AB, Buffington A, Baggett ND, Tucholka JL, Weis HB, Marka N, Schoultz T, Kalbfell E, Campbell TC, Lin V, Lape D, Brasel KJ, Phelan HA, Schwarze ML. Best case/worst case for the trauma ICU: Development and pilot testing of a communication tool for older adults with traumatic injury. J Trauma Acute Care Surg. 2021 Sep 1;91(3):542-551. doi: 10.1097/TA.0000000000003281. PMID 34039930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We received 233 survey responses for the anonymous Moral Distress Survey (MDS). As these pre/post surveys were given anonymously, it was not possible to determine the total number of participants as some participants could have completed both pre and post surveys.
Units Other Than Participants: survey responses
Groups:
- Trauma Care Provider Focus Group: Trauma Care Providers were enrolled in a focus group to assist in developing the intervention, prior to main study and randomization activities.
- Usual Care - Control Group: Usual care typically includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention. Usual care consists of daily updates with patient and family, describing each new problem as it arises and what will be done to treat it, regardless of how this fits into the patient's overall prognosis or health trajectory.
- Trauma Team Training: Using the best case/worst case training program, a trainer at the UT-S/PMH and OHSU sites trained consenting attending trauma surgeons and trauma team members. As part of the training, participants took part in an assessment session, demonstrating their use of the tool with a standardized patient and scripted clinical scenario.
- Best Case/Worst Case Communication Tool: The patient's enrolled surgeon completed training on the Best Case/Worst Case communication tool and was encouraged to use it with the patient.
  Best Case/Worst Case communication tool: The communication tool promotes dialogue and patient deliberation, and supports shared decision making in the context of life-limiting illness. Building on a conceptual model of shared decision-making proposed and the practice of scenario planning our intervention is designed to lead to a discussion of patient preferences and consideration of outcomes.
  The surgeon verbally describes the "best case," "worst case," and "most likely" outcomes for each treatment option-incorporating rich narrative from clinical experience and translation of probabilistic information-while drawing a diagram of those options. The surgeon also writes details about each option on the diagram. The narrative and graphic help family and patients formulate and express preferences.
- Participant Nurses: For the nurse-reported Quality of Communication (QoC) surveys, the primary nurse caring for an enrolled study patient was approached by a UT-S/PMH or OHSU research team member during their work shift and asked to participate by filling out a survey that assessed the QoC the patient and family have received over the prior 72 hours. Baseline characteristics were not collected for these participants and they were not randomized.
- Moral Distress Survey (MDS) Responses: All nurses and physicians of the trauma units at UT-S/PMH and OHSU were invited to participate in this brief anonymous survey given at two time points: at the start of the study before the first patient is enrolled and at the end of the study, after the last patient is enrolled. These activities occurred prior to and after the main study and randomization activities.
Period: Overall Study
Arm/Group | Trauma Care Provider Focus Group | Usual Care - Control Group | Trauma Team Training | Best Case/Worst Case Communication Tool | Participant Nurses | Moral Distress Survey (MDS) Responses
Started | 48; 0 survey responses | 48; 0 survey responses (Family members consented (24/48 had patient enroll along with them as patient had DMC).) | 62; 0 survey responses | 38; 0 survey responses (Family members consented (19/38 had patient enroll along with them as patient had DMC).) | 59; 0 survey responses | NA; 233 survey responses (Anonymous survey, cannot ascertain if same participant completed it for both pre- and post-intervention.)
Patients Who Provided Self-Consent (These participants count toward the total number of participants who 'started' the study.) | 0; 0 survey responses | 24; 0 survey responses | 0; 0 survey responses | 19; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
MDS Pre-Intervention Survey Responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 99; 99 survey responses
MDS Post-Intervention Survey Responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses | 134; 134 survey responses
Patient Survey 1 | 0; 0 survey responses | 16; 0 survey responses | 0; 0 survey responses | 13; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
Nurse Survey 1 | 0; 0 survey responses | 32; 0 survey responses | 0; 0 survey responses | 27; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
Family Survey 1 | 0; 0 survey responses | 37; 0 survey responses | 0; 0 survey responses | 38; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
Family Survey 2 | 0; 0 survey responses | 34; 0 survey responses | 0; 0 survey responses | 35; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
Family Survey 3 | 0; 0 survey responses | 29; 0 survey responses | 0; 0 survey responses | 26; 0 survey responses | 0; 0 survey responses | 0; 0 survey responses
Completed | 48; 0 survey responses | 29; 0 survey responses | 43; 0 survey responses | 26; 0 survey responses | 59; 0 survey responses | NA; 233 survey responses (Anonymous survey, cannot ascertain if same participant completed it for both pre- and post-intervention.)
Not Completed | 0; 0 survey responses | 19; 0 survey responses | 19; 0 survey responses | 12; 0 survey responses | 0; 0 survey responses | NA; 0 survey responses
Not completed — Unavailable for training | 0 | 0 | 19 | 0 | 0 | NA
Not completed — Lost to Follow-up | 0 | 18 | 0 | 11 | 0 | NA
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1 | 0 | NA

BASELINE CHARACTERISTICS:
Population: 86 family members enrolled in this study and 43 patients with decision-making capacity (DMC) associated with these family members also enrolled. Baseline characteristics are reported for the patients in both the usual care and intervention arm. For other participants, baseline characteristics were not collected and/or these participant types were not part of the study randomization schema.
Groups:
- Usual Care: Usual care typically includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention.
- Total: Total of all reporting groups
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care | Total
Number analyzed (Participants) | 38 | 48 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 0 | 8
  >=65 years | 30 | 48 | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (10.76) | 73.8 (7.25) | 73.4 (8.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 25 | 32 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 33 | 42 | 75
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 34 | 37 | 71
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 38 | 48 | 86

OUTCOME MEASURES:

1. Primary Outcome: Family Member-reported Quality of End of Life Communication (QOC) Received From Study Surgeon
Description: Family member-reported quality of end of life communication will be measured by the 7-item end of life subscale of the Quality of Communication scale. The QOC is a validated self-report instrument. The average score is given with a possible range of 0-10. Higher scores indicate higher perceived quality of end of life communication
Time Frame: 72 hours after trauma unit admission
Population: Only family members were asked to complete this survey measure (n=86). The number of participants analyzed differs from the number of total family member participants due to survey or item non-response.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Care: Usual care typically includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention. Usual care consists of daily updates with patient and family, describing each new problem as it arises and what will be done to treat it, regardless of how this fits into the patient's overall prognosis or health trajectory.
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 25 | 26
score on a scale | 6.6 (2.6) | 4.5 (2.5)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.006, t-test, 2 sided

2. Primary Outcome: Family Member-reported General Communication (QOC) Received From Study Surgeon
Description: Family member-reported general quality of end communication will be measured by the 6-item general communication subscale of the Quality of Communication scale. The QOC is a validated self-report instrument. The average score is given with a possible range of 0-10. Higher scores indicate higher perceived quality of communication
Time Frame: 72 hours after trauma unit admission
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Usual Care: Usual care typically includes informed consent and a surgeon-directed deliberative phase in which surgeons present their own evaluation of the trade-offs and goals of the proposed intervention. Usual care also consists of daily updates with patient and family, describing each new problem as it arises and what will be done to treat it, regardless of how this fits into the patient's overall prognosis or health trajectory.
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 35 | 36
score on a scale | 8.5 (1.9) | 8.3 (1.72)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.709, t-test, 2 sided

3. Secondary Outcome: Nurse-reported Quality of End of Life Communication (QOC) Received From Study Surgeon
Description: Nurse-reported quality of end of life communication will be measured by the 7-item Quality of Communication scale, end of life subscale, clinician version. The QOC is a validated self-report instrument. The average score is given with a possible range of 0-10.Higher scores indicate higher perceived quality of communication
Time Frame: 72 hours after trauma unit admission
Population: Only nurses of study patients were asked to complete this survey measure. The number of participants analyzed differs from the number of total patients (n=86) due to survey or item non-response.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 18 | 20
score on a scale | 6 (2.79) | 4.1 (2.3)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.03, t-test, 2 sided

4. Secondary Outcome: Nurse-reported General Quality of Communication (QOC) Received From Study Surgeon
Description: Nurse-reported general quality of communication will be measured by the 6-item Quality of Communication scale, general communication subscale, clinician version. The QOC is a validated self-report instrument. The average score is given with a possible range of 0-10. Higher scores indicate higher perceived quality of life communication
Time Frame: 72 hours after trauma unit admission
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 26 | 32
score on a scale | 7.7 (1.96) | 6.7 (1.97)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.063, t-test, 2 sided

5. Secondary Outcome: Family-reported Communication and Care Coordination
Description: Family-reported communication and care coordination as measured by the 30-item Family Inpatient Communication Survey (FICS). The FICS is a validated instrument. Scores on this instrument may range from 30 to 150 and higher scores indicate greater satisfaction with ICU care
Time Frame: 10 days after trauma unit admission
Population: The number of participants analyzed differs from the number of total arm participants due to a low rate of survey or item non-response. Only family members completed the 30-item Family Inpatient Communication Survey.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 35 | 33
score on a scale | 114.5 (22.98) | 113.8 (20.87)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.892, t-test, 2 sided

6. Secondary Outcome: Family-reported Goal Concordant Care
Description: Family-reported goal concordant care will be assessed by 2 survey questions taken from the SUPPORT study (Question 1: If you had to make a choice at this time, would you prefer a course of treatment for your loved one that focuses on extending life as much as possible, even if it means having more pain and discomfort, or would you want a plan of care that focuses on relieving pain and discomfort as much as possible, even if that means not living as long? Question 2: Would you say that your loved one's current medical care is more focused on extending life as much as possible, even if it means having more pain and discomfort, or on relieving pain and discomfort as much as possible, even if that means not living as long? If participant gave the same answer to both questions, this was considered to be concordant. If the answers to the 2 questions were different, this was considered discordant
Time Frame: 10 days after trauma unit admission
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 24 | 22
Participants
  Concordant | 16 | 15
  Discordant | 8 | 7
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Comparison of concordance status by intervention status (outcome by predictor); Test type: Superiority; p > . 99, Fisher Exact — Using an a priori statistical significance of 0.05

7. Secondary Outcome: Patient-reported Trauma Quality of Life (TQoL)
Description: Patient-reported trauma quality of life (TQoL) as measured by the 43 Trauma Quality of Life (TQoL) survey. The TQoL is a validated measure. Scores may range from 41-172. Higher scores indicate better quality of life
Time Frame: 30 days after trauma unit admission
Population: Only patients with decision making capacity at time of consent (n=43) were asked to complete this survey measure. The number of participants analyzed differs from the number of total patient participants due to survey or item non-response and changes in decision making capacity after consenting.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 10 | 9
score on a scale | 115.3 (17.91) | 126.7 (18.12)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.188, t-test, 2 sided

8. Secondary Outcome: Family-reported Trauma Quality of Life (TQoL)
Description: Family-reported trauma quality of life (TQoL) as measured by the 43 Trauma Quality of Life (TQoL) survey, adapted for use with family members. The TQoL is a validated measure. Scores may range from 41-172. Higher scores indicate better quality of life
Time Frame: 30 days after trauma unit admission
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 14 | 11
score on a scale | 102.6 (29.63) | 121.7 (12.56)
Statistical Analysis 1: Comparison: Best Case/Worst Case Communication Tool vs Usual Care; Test type: Superiority; p = 0.042, t-test, 2 sided

9. Secondary Outcome: Family-reported Care Quality and Bereavement
Description: Family-reported care quality and bereavement as measured by the After-Death Bereaved Family Member Interview, with questions relating to 7 domains of care quality
Time Frame: After death (in substitute for family-reported Family-reported Trauma Quality of Life)
Population: The number of participants analyzed differs from the number of total arm participants because this survey was only offered to family member participants of patients who died on study. Data was collected from 3 participants before the measure was dropped due to high participant emotional burden. Data from the 3 participants was not analyzed due to high item missingness and participant confusion and distress about survey items.
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Trauma Nurse-reported Moral Distress
Description: Trauma unit staff-reported moral distress will be measured by the 21-item Moral Distress Scale-Revised (MDS-R), nurse version. Scores many range from 0 to 336 and higher scores indicate greater moral distress
Time Frame: Start of study and 30 months after study commencement
Population: The number of participants analyzed differs from the number of total arm participants because this study activity is not associated with the registered arms; it was a pre/post instrument given at the start/end of the study to all trauma nurses present in the ICU at each of these timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention Survey: Trauma unit nurses present in the ICU will be surveyed before clinicians learn to use the best case/worst case tool (at the start of the study, before the first patient is enrolled), to assess whether the communication intervention improves feelings of moral distress.
- Post-intervention Survey: Trauma unit nurses present in the ICU will be surveyed after clinicians learn to use the best case/worst case tool (at the end of the study, after the last patient is enrolled), to assess whether the communication intervention improves feelings of moral distress.
Arm/Group | Pre-intervention Survey | Post-intervention Survey
Number analyzed (Participants) | 52 | 86
score on a scale | 79.48 (47.44) | 82.56 (40.86)
Statistical Analysis 1: Comparison: Pre-intervention Survey vs Post-intervention Survey; Test type: Superiority; p = 0.698, t-test, 2 sided

11. Secondary Outcome: Trauma Physician-reported Moral Distress
Description: Trauma unit staff-reported moral distress will be measured by the 21-item Moral Distress Scale-Revised (MDS-R), physician version. Scores many range from 0 to 336 and higher scores indicate greater moral distress
Time Frame: Start of study and 30 months after study commencement
Population: The number of participants analyzed differs from the number of total arm participants because this study activity is not associated with the registered arms; it was a pre/post instrument given at the start/end of the study to all trauma physicians present in the ICU at each of these timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-intervention Survey: Trauma physicians present in the ICU will be surveyed before clinicians learn to use the best case/worst case tool (at the start of the study, before the first patient is enrolled), to assess whether the communication intervention improves feelings of moral distress.
- Post-intervention Survey: Trauma unit physicians present in the ICU will be surveyed after clinicians learn to use the best case/worst case tool (at the end of the study, after the last patient is enrolled), to assess whether the communication intervention improves feelings of moral distress.
Arm/Group | Pre-intervention Survey | Post-intervention Survey
Number analyzed (Participants) | 38 | 36
score on a scale | 61.03 (32.32) | 51.42 (24.03)
Statistical Analysis 1: Comparison: Pre-intervention Survey vs Post-intervention Survey; Test type: Superiority; p = 0.15, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to approximately 30 days following enrollment.
Description: Participants in the pre/post moral distress surveys are not included as their participation was limited to a one-time survey. Participants in the Trauma Care Provider Focus Group, Trauma Team Training and Participant Nurses were also not formally monitored for adverse events.
Arm/Group | Best Case/Worst Case Communication Tool | Usual Care
All-Cause Mortality (participants affected / at risk) | 6/38 | 7/48
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/48
Other Adverse Events (participants affected / at risk) | 0/38 | 0/48

LIMITATIONS AND CAVEATS:
Chart-derived treatment intensity as measured by the Simplified Therapeutic Intervention Scoring System (TISS-28) was removed as an outcome measure as this data was collected inconsistently, considered unreliable and therefore not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/55/NCT03188055/Prot_SAP_000.pdf